CLINICAL TRIAL: NCT00086385
Title: Maintaining Nonsmoking: Older Smokers
Brief Title: Maintaining Nonsmoking: Older Smokers - 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIDA-02538-1; R01DA002538 (NIH); R01-02538-1
Record Dates: First submitted 2004-07-01; First posted 2004-07-07 (Estimated); Results first posted 2013-10-10 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2015-03

CONDITIONS: Tobacco Use Disorder
Keywords: Smoking cessation; Tobacco
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation | interventions — Tobacco Use Cessation Devices; Bupropion; Nicotine Chewing Gum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Brief Treatment (Active Comparator): Pharmacological Treatment - Subjects received 12 weeks of bupropion treatment and 10 weeks of nicotine replacement treatment (NRT)
  Brief Counseling - The counseling intervention consisted of five 90-minute group meetings.
  There was no further treatment during Weeks 12-52.
  Interventions: Drug: Nicotine polacrilex, Bupropion
- Extended NRT (Experimental): Pharmacological Treatment - Following completion of the Brief Treatment, subjects assigned to this condition would continue receiving NRT for up to 52 weeks. Subjects in this condition would be encouraged to continue NRT through Week 24. If a subject terminated NRT and resumed smoking, before Week 50, would be instructed to set a quit date and resume NRT.
  Counseling Treatment - This is identical to the Brief Counseling described above.
  Interventions: Drug: Nicotine polacrilex, Bupropion
- Tailored/No Extended NRT (Experimental): This condition was identical to the Tailored/NRT condition except that no NRT was available after completion of the Brief Treatment.
  Interventions: Drug: Nicotine polacrilex, Bupropion
- Extended Tailored Counseling + NRT (Experimental): Tailored Counseling Treatment- The primary goal of the extended treatment was to prevent relapse. Secondary goal was to encourage initiation of abstinence for those who have not attained it by Week 12, and re-initiation of abstinence after slips. Subjects would participate in the Brief Treatment followed by individual sessions. The first extended treatment counseling session would occur at Week 10. Additional sessions would be held every two weeks then every four weeks, and finally at Weeks 44 and 52. Each session would be 20-30 minutes long. Between sessions subjects would be contacted by phone for brief check-ins (5-10 minutes).
  Interventions: Drug: Nicotine polacrilex, Bupropion

INTERVENTIONS:
Drug: Nicotine polacrilex, Bupropion — Subjects receive 12 weeks of bupropion treatment and 10 weeks of nicotine replacement.
  Other Names: Nicorette, Zyban

SUMMARY:
The purpose of this study was to examine pharmacological and psychological interventions for smokers over 50.

DETAILED DESCRIPTION:
The overall goals of this line of research were to prevent relapse to cigarette smoking, and to understand the processes related to smoking and relapse. The specific aims of the current study were to test a series of hypotheses about the efficacy and cost-effectiveness of long-term, tailored interventions in chronic, older smokers and the interaction of these interventions with gender and depression. Participants were 50 years or older and smoker 10 or more cigarettes per day. Baseline assessments includes measures of smoking behavior, nicotine dependence, depression diagnosis, demographics and life circumstances and measures of anger, depression and mood disturbance, stress, social support, health status, motivation for changed and drug and alcohol use.

ELIGIBILITY:
smokers of at least 10 cigarettes per day

Inclusion Criteria:

MULTIPLE

Exclusion Criteria:

MULTIPLE

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 403 (Actual)
Dates: Start 2001-09; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon M Hall, Ph.D., Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco, San Francisco, California, United States

REFERENCES:
- [Derived] Theodoulou A, Fanshawe TR, Leavens E, Theodoulou E, Wu AD, Heath L, Stewart C, Nollen N, Ahluwalia JS, Butler AR, Hajizadeh A, Thomas J, Lindson N, Hartmann-Boyce J. Differences in the effectiveness of individual-level smoking cessation interventions by socioeconomic status. Cochrane Database Syst Rev. 2025 Jan 27;1(1):CD015120. doi: 10.1002/14651858.CD015120.pub2. PMID 39868569
- [Derived] Theodoulou A, Chepkin SC, Ye W, Fanshawe TR, Bullen C, Hartmann-Boyce J, Livingstone-Banks J, Hajizadeh A, Lindson N. Different doses, durations and modes of delivery of nicotine replacement therapy for smoking cessation. Cochrane Database Syst Rev. 2023 Jun 19;6(6):CD013308. doi: 10.1002/14651858.CD013308.pub2. PMID 37335995
- [Derived] Barnett PG, Wong W, Jeffers A, Munoz R, Humfleet G, Hall S. Cost-effectiveness of extended cessation treatment for older smokers. Addiction. 2014 Feb;109(2):314-22. doi: 10.1111/add.12404. Epub 2013 Dec 13. PMID 24329972
- [Derived] Hall SM, Humfleet GL, Munoz RF, Reus VI, Robbins JA, Prochaska JJ. Extended treatment of older cigarette smokers. Addiction. 2009 Jun;104(6):1043-52. doi: 10.1111/j.1360-0443.2009.02548.x. Epub 2009 Apr 9. PMID 19392908

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects will be men and women, 50 years and older who smoke at least 10 cigarettes a day. They will respond to requests in the public media for individuals who are interested in quitting smoking, and will be referred from sources like UCSF Ambulatory Care Clinics, California Pacific General Medical Practice, and Jewish Family and Community Center.
Pre-assignment Details: One participant died at week 5 before randomization.
Groups:
- Brief Treatment: Pharmacological Treatment - Subjects receive 12 weeks of bupropion treatment and 10 weeks of nicotine replacement treatment
  Brief Counseling - The counseling intervention consist of five 90-minute group meetings.
  No further treatment during Weeks 12-52.
  Nicotine polacrilex, Bupropion : Subjects receive 12 weeks of bupropion treatment and 10 weeks of nicotine replacement.
- Extended NRT: Pharmacological Treatment - Following completion of the Brief Treatment, subjects assigned to this condition will continue receiving NRT for up to 52 weeks. Subjects in this condition will be encouraged to continue NRT through Week 24. If a subject who terminates NRT and resumes smoking, before Week 50, will be instructed to set a quite date and resume NRT.
  Counseling Treatment - This is identical to the Brief Counseling described above.
  Nicotine polacrilex, Bupropion : Subjects receive 12 weeks of bupropion treatment and 10 weeks of nicotine replacement.
- Extended Tailored Counseling + NRT: Tailored Counseling Treatment- The primary goal of the extended treatment is to prevent relapse. Secondary goal is to encourage initiation of abstinence for those who have no attained it by Week 12, and re-initiation of abstinence after slips. Subjects will participate in the Brief Treatment followed by individual sessions. The first extended treatment counseling session will occur at Week 10. Additional sessions will be held every two weeks then every four weeks, and finally at Weeks 44 and 52. Each session will be 20-30 minutes long. Between sessions subjects will be contacted by phone for brief check-ins (5-10 minutes).
  Nicotine polacrilex, Bupropion : Subjects receive 12 weeks of bupropion treatment and 10 weeks of nicotine replacement.
- Tailored/No Extended NRT: This condition is identical to the Tailored/NRT condition except that no NRT is available after completion of the Brief Treatment.
  Nicotine polacrilex, Bupropion : Subjects receive 12 weeks of bupropion treatment and 10 weeks of nicotine replacement.
Period: Overall Study
Arm/Group | Brief Treatment | Extended NRT | Extended Tailored Counseling + NRT | Tailored/No Extended NRT
Started | 100 | 99 | 104 | 99
Completed | 98 | 97 | 103 | 98
Not Completed | 2 | 2 | 1 | 1
Not completed — Death | 2 | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brief Treatment | Extended NRT | Extended Tailored Counseling + NRT | Tailored/No Extended NRT | Total
Number analyzed (Participants) | 100 | 99 | 104 | 99 | 402
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 93 | 86 | 94 | 85 | 358
  >=65 years | 7 | 13 | 10 | 14 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.190 (5.40) | 56.97 (5.46) | 56.88 (6.82) | 56.63 (5.64) | 56.67 (5.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 40 | 39 | 41 | 161
  Male | 59 | 59 | 65 | 58 | 241
Region of Enrollment [Number; unit: participants]
  United States | 100 | 99 | 104 | 99 | 402

OUTCOME MEASURES:

1. Primary Outcome: Participants Abstinent From Cigarettes
Description: Primary outcome variable was 7-day point prevalence cigarette abstinence verified biochemically at week 104
Time Frame: Two years
Measure: Number; unit: participants
Arm/Group | Brief Treatment | Extended NRT | Extended Tailored Counseling + NRT | Tailored/No Extended NRT
Number analyzed (Participants) | 100 | 99 | 104 | 99
participants | 31 (5.4) | 35 (6.82) | 39 (5.64) | 45 (5.46)

ADVERSE EVENTS:
Time Frame: Baseline to week 104.
Arm/Group | Brief Treatment | Extended NRT | Extended Tailored Counseling + NRT | Tailored/No Extended NRT
Serious Adverse Events (participants affected / at risk) | 2/100 | 5/99 | 4/104 | 2/99
Other Adverse Events (participants affected / at risk) | 1/100 | 3/99 | 4/104 | 3/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brief Treatment (N=100) | Extended NRT (N=99) | Extended Tailored Counseling + NRT (N=104) | Tailored/No Extended NRT (N=99)
Death (not related to study) (General disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (1) — Ruled unrelated serious adverse event.
Angina (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Ruled unrelated serious adverse event to the study. Hospitalized.
Heart Procedure (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Ruled unrelated serious adverse event. Hospitalized for a heart procedure.
Implantation of an Automatic Implantable Cardioverter Defibrillator (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Ruled unrelated serious adverse event. Hospitalized.
Asthma Attack (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Reported unrelated serious adverse event. Hospitalized.
Myocardial Infarct (MI) (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Reported unrelated serious adverse event. Hospitalized.
Fatigue, Weakness, and Unsteady Walking (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Reported unrelated serious adverse event. Hospitalized.
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Ruled unrelated serious adverse event. Hospitalized.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brief Treatment (N=100) | Extended NRT (N=99) | Extended Tailored Counseling + NRT (N=104) | Tailored/No Extended NRT (N=99)
Lung Biopsy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Ruled unrelated adverse event.
Midsternal Pressure (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Ruled directly related adverse event. Her blood pressure and heart rate were ruled normal by the study's staff. Subject was advise to discontinue gum use and seek appt with primary care provider.
Anxiety, High Blood Presure (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Ruled indirectly related adverse event. Subject discontinued study medication.
Dental Issues (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) — Ruled unrelated adverse event.
Insomnia (General disorders) | 0 (0) | 1 (2) | 1 (1) | 2 (2) — Ruled unrelated adverse event.
Numbness/Tingling (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Ruled unrelated adverse event.

LIMITATIONS AND CAVEATS:
The limitations of this study include generalizability, as the population treated was relatively well-educated, willing to participate in research and to attend treatment sessions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No